CLINICAL TRIAL: NCT02109276
Title: Contrast Sensitivity and Higher Order Aberrations After Spheric and Aspheric Intraocular Lens Implantation for Patients With Mild to Moderate Fuch's Endothelial Dystrophy.
Brief Title: Study of the Effect of Aspheric Lenses in Patients With Fuch's Dystrophy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough participants
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Stephanie Baxter, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPTH-151-14
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Fuch's Endothelial Dystrophy; Cataracts
Keywords: Fuch's endothelial dystrophy; Aspheric intraocular lens; Higher Order Aberrations; Contrast Sensitivity
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spheric Sensar(R) 3-piece IOL (Active Comparator): This group of patients with Fuchs endothelial dystrophy and cataract will undergo cataract extraction and be randomized to receive a Spheric Sensar(R) 3-piece IOL
  Interventions: Device: Spheric Sensar(R) 3-piece IOL
- Aspheric Tecnis(R) 3-piece IOL (Experimental): This group of patients with Fuchs endothelial dystrophy and cataract will undergo cataract extraction and be randomized to receive an Aspheric Tecnis(R) 3-piece IOL
  Interventions: Device: Aspheric Tecnis(R) 3-piece IOL

INTERVENTIONS:
Device: Spheric Sensar(R) 3-piece IOL — Patients will be randomized to receive either a standard spheric intraocular lens or an aspheric intraocular lens
  Arms: Spheric Sensar(R) 3-piece IOL
Device: Aspheric Tecnis(R) 3-piece IOL — Patients will be randomized to receive either a standard spheric intraocular lens or an aspheric intraocular lens
  Arms: Aspheric Tecnis(R) 3-piece IOL

SUMMARY:
The proposed study will recruit patients with mild to moderate Fuch's dystrophy who need cataract surgery alone. They will be randomly assigned to receive either spheric or aspheric lenses. If both eyes of a patient need surgery, we will implant the same type of lens in each eye in order to prevent imbalanced vision. We will measure their contrast sensitivity and higher order aberrations before surgery and 3 months after surgery. We will compare the change in these values between the two groups.

DETAILED DESCRIPTION:
Fuch's endothelial dystrophy is a disease of the human cornea, which affects people in the fifth or sixth decade of life. Due to poorly functioning cells its inner surface, the cornea becomes swollen, resulting in pain and blurry vision. Mild to moderate Fuch's disease can be managed pharmacologically or conservatively. Nonetheless, cataract development is an unrelated age-associated process that occurs in the same way in patients with and without Fuch's endothelial dystrophy. Therefore, many patients with mild to moderate Fuch's dystrophy would need to undergo cataract surgery.

In cataract surgery, the native human lens is removed and replaced with a synthetic intraocular lens. There are several varieties of lenses available currently. Of these, the aspheric lens has a unique contour that was developed to complement the surface features of the cornea, thus reducing spherical aberrations. Several studies have shown that the aspheric lens improves contrast sensitivity in dim light and higher order aberrations in the otherwise normal eye. Contrast sensitivity refers to the ability of the patient to discern differences in similar shades of colour. Higher order aberration is a concept that is used to quantify how much the optical mechanism of the eye distorts incoming light rays. Most of these studies compared the aspheric lens to the standard spheric lens.

Since Fuch's patients can experience intermittent corneal swelling, the shape of their corneal surface is prone to distortion. Since the aspheric lens does not change shape, it is unknown how its fixed surface will interact with the fluctuating corneal surface in patients with Fuch's endothelial dystrophy.

To date, there have been no studies looking at contrast sensitivity and higher order aberrations in patients with Fuch's dystrophy who were implanted with an aspheric intraocular lens. The accepted practice is to offer Fuch's patients the aspheric lens during the pre-operative evaluation, and explain to them that we are not sure how it will be of benefit to them. At Hotel Dieu Hospital in Kingston, there is a cost of $125 to all patients who choose the aspheric lens, while the spheric lens is free. Therefore, most patients with Fuch's dystrophy choose the spheric lens. There is no evidence-based data to guide patient choice in this situation.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and 80 years
* Visual acuity better than 0.2 logMAR units
* preoperative corneal spherical aberration (Zo4) values between 0.1 and 0.25 µm at 5-mm pupil diameter
* IOL power between +18.00 and +24.00 diopters

Exclusion Criteria:

* Intraocular lens tilt and decentration estimated by retroillumination
* surgical complications
* posterior capsule rupture
* residual posterior capsule plaque
* posterior capsular opacity
* post operative Best Corrected Visual Acuity <20/25
* corneal astigmatism >= 1.00 D
* glaucoma
* amblyopia,
* history of uveitis
* diabetic retinopathy,
* pseudoexfoliation syndrome
* macular pathology previous intraocular surgery
* coexisting ocular pathology
* axial length >25mm
* non dilating pupils
* corneal laser therapy
* poor follow up
* use of topical medications (apart from lubricants)
* systemic steroids use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in contrast sensitivity. | 3 months (plus or minus 1 week) post operatively

SECONDARY OUTCOMES:
Higher Order Aberrations | 3 months (plus or minus 1 week) post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Baxter, MD, FRCSC, Principal Investigator — Department of Ophthalmology, Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada